CLINICAL TRIAL: NCT00501293
Title: A Phase IIIb, Long-Term, Open-Label, Multi-Center, Extension Study Designed to Evaluate the Safety and Efficacy of Methylphenidate Transdermal System (MTS) in Adolescents Aged 13-17 Years With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Evaluate the Safety and Efficacy of Methylphenidate Transdermal System (MTS) in Adolescents Aged 13-17 Years With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD485-410
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Results first posted 2010-01-15 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Methylphenidate Transdermal System
  Interventions: Drug: Methylphenidate Transdermal System

INTERVENTIONS:
Drug: Methylphenidate Transdermal System — One of 4 doses of the MTS transdermal patch over the same duration of wear for approximately 6 months
  Other Names: DAYTRANA

SUMMARY:
To evaluate the long-term, safety of Methylphenidate Transdermal System (MTS) in aged 13-17 years diagnosed withADHD

DETAILED DESCRIPTION:
To evaluate the long-term, safety of Methylphenidate Transdermal System (MTS) in the symptomatic treatment of adolescents aged 13-17 years diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD) by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria. The evaluation of safety will be based on treatment-emergent adverse events (TEAEs), laboratory tests, vital signs, physical examinations, electrocardiograms (ECGs), and skin tolerability to MTS based on the dermal response score (DRS).

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, each subject must fulfill each of the following criteria at the Entry visit:

* The subject participated in the antecedent SPD485-409 study, and a) completed all required study visits (Baseline through Visit 9) OR b) completed the 5 week Dose Optimization period without achieving an acceptable condition as defined by the antecedent SPD485-409 study.
* Subject has blood pressure measurements within the 95th percentile for age, gender, and height at Entry.
* Subject's ECG results are within the normal range or not clinically significant at Entry as judged by the Investigator in conjunction with the central reader.
* Females must have a negative urine pregnancy test at Entry and agree to use acceptable contraceptives throughout the study period and for 30 days the last dose of IP.
* Subject and parent of legally authorized representative (LAR) are able, willing and likely to fully comply with study procedures and restrictions.
* Written, signed and dated informed consent to participate in the study must be given by the subject's parent or LAR, in accordance with the International Conference on Harmonisation (ICH), Good Clinical Practices (GCP) Guideline E6 and applicable regulations, before completing any study-related procedures.
* There must be documentation of the subject's assent to participate in the study indicating that the subject is aware of the investigational nature of the study and the required procedures and restrictions. Failure to object is not to be considered assent.

Exclusion Criteria

Subjects will be excluded from the study if any of the following criteria are met at Entry:

* Subject was discontinued from SPD485-409 due to a protocol violation, non-compliance, AE, or a serious adverse event (SAE).
* Subject has a concurrent chronic or acute illness (such as severe allergic rhinitis or an infectious process requiring antibiotics), disability, or other condition that might confound the results of safety assessments administered in the study or that might increase risk to the subject. Similarly, the subject will be excluded if he or she has any additional condition(s) that in the Investigator's opinion would prohibit the subject from completing the study or would not be in the best interest of the subject. This would include any significant illness or unstable medical condition that could lead to difficulty complying with the protocol. Mild, stable asthma is not exclusionary.
* Subject is taking any medication that is excluded.
* Female subject who is pregnant or lactating.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Findling, M.D., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (32):
- United States (32):
  - Melmed Center, Scottsdale, Arizona
  - Bay Area Research Institute, Lafayette, California
  - Elite Clinical Trials Inc., Wildomar, California
  - Sarkis Clinical Trials, Gainsville, Florida
  - Miami Research Associates, South Miami, Florida
  - Northwest Behavioral Research Ctr, Roswell, Georgia
  - Mountain West Clinical Trials, LLC, Eagle, Idaho
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Shire Clinical Research Site, Lexington, Kentucky
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Clinical Neurophysiology Services, PC, Troy, Michigan
  - CRI Worldwide, Clementon, New Jersey
  - Triangle Neuropsychiatry, Durham, North Carolina
  - Dakota Clinic/Innovis Health, Fargo, North Dakota
  - Odyssey Research, Minot, North Dakota
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Oregon center for Clinical Investigations, Inc., Eugene, Oregon
  - OCCI, Inc, Portland, Oregon
  - Shire Clinical Research Site, Media, Pennsylvania
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - CNS Healthcare, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Claghorn-Lesem Research, Ltd., Bellaire, Texas
  - Westex Clinical Investigations, Lubbock, Texas
  - Cerebral Research, LLC, San Antonio, Texas
  - Vermont Clinical Study Center, Burlington, Vermont
  - NeuroScience, Inc., Herndon, Virginia
  - Adolescent Health Center, Midlothian, Virginia
  - Northwest Clinical Research Center, Friday Harbor, Washington
  - Eastside Therapeutic Resource, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Findling RL, Katic A, Rubin R, Moon E, Civil R, Li Y. A 6-month, open-label, extension study of the tolerability and effectiveness of the methylphenidate transdermal system in adolescents diagnosed with attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2010 Oct;20(5):365-75. doi: 10.1089/cap.2009.0122. PMID 20973707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, extension study of Methylphenidate Transdermal System (MTS) in subjects who had previously received study medication (MTS or placebo) in the antecedent study, SPD485-409 (NCT00499863). Upon entry into this study (SPD485-410), all subjects received MTS treatment regardless of the study treatment they had received in study SPD485-409.
Pre-assignment Details: The study consisted of a dose optimization period (approx. 5 weeks) and a maintenance period (5 months). Methylphenidate Transdermal System (MTS)(10, 15, 20 or 30 mg / 9 hour dose patch) was applied once-daily on the alternating hip for a 9-hour wear time. One subject in the MTS group was enrolled in error and was removed prior to receiving drug.
Groups:
- Antecedent Methylphenidate Transdermal System (MTS): Subjects who had previously received MTS in the antecedent study, SPD485-409. Upon entry into this study (SPD485-410), all subjects received MTS treatment.
- Antecedent Placebo: Subjects who had previously received placebo in the antecedent study, SPD485-409. Upon entry into this study (SPD485-410), all subjects received MTS treatment.
Period: Optimization Period
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Started | 110 | 53
Completed | 109 | 53
Not Completed | 1 | 0
Not completed — Enrolled in error | 1 | 0
Period: Maintenance Period
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Started | 109 | 53
Completed | 63 | 25
Not Completed | 46 | 28
Not completed — Withdrawal by Subject | 14 | 13
Not completed — Lost to Follow-up | 12 | 7
Not completed — Adverse Event | 6 | 6
Not completed — Protocol Violation | 2 | 1
Not completed — Lack of Efficacy | 4 | 1
Not completed — Noncompliant with study medication | 5 | 0
Not completed — Went into rehabilitation | 1 | 0
Not completed — Would not wear patch | 1 | 0
Not completed — Application site reaction | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo | Total
Number analyzed (Participants) | 110 | 53 | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 110 | 53 | 163
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (1.18) | 14.5 (1.37) | 14.5 (1.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 14 | 41
  Male | 83 | 39 | 122
Region of Enrollment [Number; unit: participants]
  United States | 110 | 53 | 163

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale-fourth Edition (ADHD-RS-IV) Scores at 6 Months
Description: The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and 6 months
Population: Intent-to-treat (ITT) defined as subjects who were enrolled and received at least one dose of MTS and had at least one assessment of the primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Number analyzed (Participants) | 106 | 52
Units on a scale
  Baseline measure | 16.0 (12.00) | 27.4 (12.91)
  6 months | 13.5 (10.55) | 14.5 (9.53)
  Change from baseline at 6 months | -2.6 (11.80) | -12.9 (15.20)
Statistical Analysis 1: Comparison: Antecedent Methylphenidate Transdermal System (MTS); Test type: Superiority or Other; p = 0.028, t-test, 2 sided; t-test of MTS at baseline and 6 months
Statistical Analysis 2: Comparison: Antecedent Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; t-test of placebo at baseline and 6 months

2. Secondary Outcome: Change From Baseline in Conner's Parent Rating Scale-revised Short Version (CPRS-R) at 6 Months
Description: The Conner's Parent rating Scale-revised short version (CPRS-R) consists of 27 questions graded on a scale from 0 (not true at all) to 3 (very much true) with a total score ranging from 0 to 81. Higher scores are indicative of increased ADHD. This scale allows parents to respond on the basis of the child's behavior and help assess ADHD and evaluate problem behavior.
Time Frame: Baseline and 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Number analyzed (Participants) | 105 | 52
Units on a scale
  Baseline measure | 26.5 (18.22) | 42.3 (16.94)
  6 months | 22.5 (16.68) | 24.6 (12.92)
  Change from baseline at 6 months | -3.9 (17.91) | -17.7 (20.10)
Statistical Analysis 1: Comparison: Antecedent Methylphenidate Transdermal System (MTS); Test type: Superiority or Other; p = 0.027, t-test, 2 sided; t-test of MTS at baseline and 6 months
Statistical Analysis 2: Comparison: Antecedent Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; t-test of placebo at baseline and 6 months

3. Secondary Outcome: Number of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) Scores
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 6 months
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Number analyzed (Participants) | 106 | 52
Participants | 81 | 39

4. Secondary Outcome: Number of Participants With Improvement on Parent Global Assessment (PGA) Scores.
Description: Parent Global Assessment (PGA) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 6 months
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Number analyzed (Participants) | 106 | 52
Participants | 69 | 31

5. Secondary Outcome: Change From Baseline in Youth Quality of Life-research Version (YQOL-R) Total Score at 6 Months
Description: The Youth Quality of Life-research version (YQOL-R) is a validated 56-item generic instrument for comparing quality of life of adolescents across condition groups that scores each question on a scale from 0 (never) to 4 (very often). The YQOL scores are transformed to a 0-100 scale for easy interpretability. Higher scores indicate better quality of life.
Time Frame: Baseline and 6 months
Population: ITT. Not all subjects in the ITT population completed a YQOL-R.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Number analyzed (Participants) | 84 | 33
Units on a scale
  Baseline measure | 82.4 (14.28) | 80.9 (14.61)
  6 months | 85.0 (13.00) | 84.6 (10.78)
  Change from baseline at 6 months | 1.9 (9.57) | 2.7 (6.23)
Statistical Analysis 1: Comparison: Antecedent Methylphenidate Transdermal System (MTS); Test type: Superiority or Other; p = 0.071, t-test, 2 sided; t-test of MTS at baseline and 6 months
Statistical Analysis 2: Comparison: Antecedent Placebo; Test type: Superiority or Other; p = 0.017, t-test, 2 sided; t-test of placebo at baseline and 6 months

6. Primary Outcome: Systolic Blood Pressure
Time Frame: Baseline and 6 months
Population: Safety population defined as all subjects that received at least one dose of MTS.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Number analyzed (Participants) | 109 | 53
mmHg
  Baseline measure | 113.4 (9.59) | 113.0 (11.20)
  6 months | 115.3 (9.91) | 115.9 (14.82)

7. Primary Outcome: Diastolic Blood Pressure
Time Frame: Baseline and 6 months
Population: Safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Number analyzed (Participants) | 109 | 53
mmHg
  Baseline measure | 69.4 (7.42) | 67.2 (7.69)
  6 months | 67.9 (7.79) | 68.9 (8.28)

8. Primary Outcome: Pulse Rate
Time Frame: Baseline and 6 months
Population: Safety population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Number analyzed (Participants) | 109 | 53
beats per minute
  Baseline measure | 80.4 (11.34) | 74.3 (9.73)
  6 months | 81.7 (11.60) | 78.9 (12.27)

9. Primary Outcome: Electrocardiogram Results (QTcF Interval)
Description: QTcF is the QT interval using Fridericia's correction formula. QT interval is a measure of time between the start of the Q wave and the end of the T wave and is dependent on the heart rate(e.g., the faster the heart rate, the shorter the QT interval). The QT interval has to be corrected in order to aid interpretation.
Time Frame: Baseline and 6 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Number analyzed (Participants) | 108 | 52
msec
  Baseline measure | 391.8 (20.76) | 393.2 (17.85)
  6 months | 395.3 (21.22) | 393.5 (21.53)

10. Primary Outcome: Post Sleep Questionnaire (PSQ) Quality of Sleep
Description: Post Sleep Questionnaire (PSQ) overall rating of quality of sleep. There are 5 rating responses ranging from very poor to very good. No numbers are associated with the rating responses.
Time Frame: 6 months
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Number analyzed (Participants) | 91 | 38
Participants
  Very poor | 1 | 1
  Poor | 6 | 3
  Average | 34 | 10
  Good | 27 | 15
  Very Good | 23 | 9

11. Primary Outcome: Weight
Time Frame: Baseline and 6 months
Population: Safety population
Measure: Mean (Standard Deviation); unit: lb
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Number analyzed (Participants) | 109 | 53
lb
  Baseline measure | 127.05 (24.003) | 131.95 (29.862)
  6 months | 134.55 (25.575) | 124.78 (29.083)

12. Primary Outcome: Dermal Reactions
Description: Dermal reactions were graded on a scale ranging from 0 (no irritation) to 7 (strong reaction) for observed findings of erythema, edema, papules, and vesicles.
Time Frame: 6 months
Population: Safety Population
Measure: Number; unit: Participants
Groups:
- Antecedent MTS and Antecedent Placebo: Methylphenidate Transdermal System and Placebo Patch
Arm/Group | Antecedent MTS and Antecedent Placebo
Number analyzed (Participants) | 162
Participants
  0 (No evidence of irritation) | 23
  1 (Minimal erythema) | 42
  2 (Definite erythema) | 82
  3 (Erythema and papules) | 6
  4 (Definite edema) | 0
  5 (Erythema, edema, and papules) | 4
  6 (Vesicular eruption) | 0
  7 (Strong reaction beyond test site) | 0
  No dermal evaluation | 5

ADVERSE EVENTS:
Description: Safety population defined as all subjects who received at least one dose of MTS.
Arm/Group | Antecedent Methylphenidate Transdermal System (MTS) | Antecedent Placebo
Serious Adverse Events (participants affected / at risk) | 3/109 | 1/53
Other Adverse Events (participants affected / at risk) | 36/109 | 32/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antecedent Methylphenidate Transdermal System (MTS) (N=109) | Antecedent Placebo (N=53)
Seizure (Nervous system disorders) | 2 | 0
Hallucinations (Psychiatric disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antecedent Methylphenidate Transdermal System (MTS) (N=109) | Antecedent Placebo (N=53)
Nasopharyngitis (Infections and infestations) | 10 | 3
Upper respiratory tract infection (Infections and infestations) | 11 | 6
Decreased appetite (Metabolism and nutrition disorders) | 12 | 13
Headache (Nervous system disorders) | 11 | 8
Irritability (Psychiatric disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.